CLINICAL TRIAL: NCT01157286
Title: Obstructive Apnea in Patients Submitted to Partial Laryngectomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital do Servidor Publico Estadual (Other)
Responsible Party: Raquel Chartuni Pereira Teixeira, resident
Other Study IDs: SAOS1
Record Dates: First submitted 2010-07-06; First posted 2010-07-07 (Estimated); Last update posted 2018-03-12 (Actual); Status verified 2010-07

CONDITIONS: OBSTRUCTIVE SLEEP APNEA
Keywords: OBSTRUCTIVE SLEEP APNEA LARINGECTOMY CPAP
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- level of apnea: patients will be separated depending on the iah(apnea hypopnea index) in mild, moderate and severe

SUMMARY:
The investigators intend to study the prevalence of obstructive apnea in patients submitted to partial laryngectomy by larynx cancer. Volunteers will be evaluated using polissonografy. We will try to correlate the residual glotic area with the number of apneas per hour.

DETAILED DESCRIPTION:
We are trying to avaliate the residual glotic area using spirometry e laryngoscopy

ELIGIBILITY:
Inclusion Criteria:

* PARTIAL LARINGECTOMY, OVER 18 YEARS,

Exclusion Criteria:

* TRACHEOSTOMY DEPRESSION USE OF DRUGS SEVERE DPOC CANCER RECURRENCE

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PATIENTS OVER 18 YEARS, SUBMITED IN THE LAST 15 YEARS TO PARTIAL LARINGECTOMY IFNO TRACHEOSTOMY IS PRESENT
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2010-06; Primary Completion 2011-07 (Estimated); Study Completion 2011-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: raquel teixeira, doctor, Principal Investigator — HSPE; Raquel Teixeira, doctor, Principal Investigator — pos graduatin student
Locations (1):
- Instituto de Assistência Médica ao Servidor Público Estadual, São Paulo, Brazil